CLINICAL TRIAL: NCT02737475
Title: A Phase 1/2a Study of BMS-986178 Administered Alone or in Combination With Nivolumab and/or Ipilimumab in Subjects With Advanced Solid Tumors
Brief Title: An Investigational Immuno-Therapy Study of Experimental Medication BMS-986178 by Itself or in Combination With Nivolumab and/or Ipilimumab in Participants With Solid Cancers That Are Advanced or Have Spread
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA012-004; 2015-004816-39 (EudraCT Number)
Record Dates: First submitted 2016-04-08; First posted 2016-04-14 (Estimated); Results first posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Nivolumab; Ipilimumab; Tetanus Toxoid; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1: Dose Escalation (Experimental): * BMS-986178 at specified doses at specified intervals
  * Enrollment is closed for this arm
  Interventions: Drug: BMS-986178
- Part 2: Dose Escalation and Expansion (Experimental): * BMS-986178 in combination with Nivolumab at specified doses at specified intervals
  * Enrollment is closed for this arm
  Interventions: Drug: BMS-986178; Drug: Nivolumab
- Part 3: Dose Escalation and Expansion (Experimental): * BMS-986178 in combination with Ipilimumab at specified doses at specified intervals
  * Enrollment is closed for this arm
  Interventions: Drug: BMS-986178; Drug: Ipilimumab
- Part 4: Dose Schedule and Exploration (Experimental): * BMS-986178/Nivolumab at specified doses at specified intervals
  * Enrollment is closed for this arm
  Interventions: Drug: BMS-986178; Drug: Nivolumab
- Part 5: Dose Schedule and Exploration (Experimental): * BMS-986178/Ipilimumab at specified doses at specified intervals
  * Enrollment is closed for this arm
  Interventions: Drug: BMS-986178; Drug: Ipilimumab
- Part 6: Dose Safety and Expansion (Experimental): * BMS-986178/Ipilimumab/Nivolumab at specified doses at specified intervals
  * Enrollment is closed for this arm
  Interventions: Drug: BMS-986178; Drug: Nivolumab; Drug: Ipilimumab
- Part 7: Dose Safety and Expansion (Experimental): * BMS-986178/Ipilimumab/Nivolumab at specified doses at specified intervals
  * Enrollment is closed for this arm
  Interventions: Drug: BMS-986178; Drug: Nivolumab; Drug: Ipilimumab
- Part 8: Dose Exploration (Experimental): * BMS-986178/Nivolumab with tetanus vaccine at specified doses and interval
  * Enrollment is closed for this arm
  Interventions: Drug: BMS-986178; Drug: Nivolumab; Biological: Tetanus vaccine
- Part 9: Dose Exploration (Experimental): * BMS-986178/Nivolumab/DPV-001 vaccine/cyclophosphamide (cohort 1) at specified doses at specified intervals OR Nivolumab/DPV-001 vaccine/cyclophosphamide (cohort 2) at specified doses at specified intervals
  * Enrollment is open for this arm [Tumor type triple negative breast cancer (TNBC)]
  Interventions: Drug: BMS-986178; Drug: Nivolumab; Biological: DPV-001 vaccine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: BMS-986178 — Specified dose on specified days
Drug: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
  Arms: Part 2: Dose Escalation and Expansion; Part 4: Dose Schedule and Exploration; Part 6: Dose Safety and Expansion; Part 7: Dose Safety and Expansion; Part 8: Dose Exploration; Part 9: Dose Exploration
Drug: Ipilimumab — Specified dose on specified days
  Other Names: BMS-734016; Yervoy
  Arms: Part 3: Dose Escalation and Expansion; Part 5: Dose Schedule and Exploration; Part 6: Dose Safety and Expansion; Part 7: Dose Safety and Expansion
Biological: Tetanus vaccine — Specified dose on specified days
  Arms: Part 8: Dose Exploration
Biological: DPV-001 vaccine — DPV-001 (UbiLT3 and UbiLT6): Specified dose on specified days
  Arms: Part 9: Dose Exploration
Drug: Cyclophosphamide — Specified dose on specified days
  Arms: Part 9: Dose Exploration

SUMMARY:
The purpose of the study is to determine the safety and tumor-shrinking ability of experimental medication BMS-986178, when given by itself or in combination with Nivolumab and/or Ipilimumab, in participants with solid cancers that are advanced or have spread.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

For Part 9 (only arm open for enrollment):

* Stage IV metastatic or unresectable triple negative breast cancer (TNBC) with zero or one prior systemic therapies in the advanced metastatic setting
* Participants with < 12 months from receipt of last curative-intent chemotherapy are allowed; curative chemotherapy will be considered first-line therapy
* Prior receipt of chemotherapy in the (neo)adjuvant setting is acceptable, as long as completed greater than 6 months from start of treatment
* Tumor biopsy samples (mandatory pre- and on-treatment biopsies) are required for all participants enrolled
* Must have histologic or cytologic confirmation of a malignancy that is advanced (metastatic, recurrent, refractory, and/or unresectable) with measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
* Men and women must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Must be immunotherapy treatment naïve, including no prior therapy with T cell immune checkpoint blocker (anti-PDL1, anti-PD1). Prior receipt of intralymphatic cytokine therapy (IRX-2) is acceptable (Part 9 only)
* Other active malignancy requiring concurrent intervention
* Prior therapy with any agent specifically targeting T-cell co-stimulation pathways such as anti-OX40 antibody, anti-CD137, anti- glucocorticoid-induced TNFR-related gene (anti-GITR) antibody, and anti-CD27
* Known or underlying medical or psychiatric condition and/or social reason that, in the opinion of the investigator or Sponsor, could make the administration of study drug hazardous to the participant or could adversely affect the ability of the participant to comply with or tolerate the study

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2016-06-17 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (22):
- United States (8):
  - University Of Colorado, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center (Cumc), New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario
- Israel (2):
  - Local Institution, Ramat Gan
  - Local Institution, Tel Aviv
- Italy (2):
  - IRCCS Istituto Nazionale Tumori Milano, Milan
  - Istituto Clinico Humanitas, Rozzano
- Netherlands (2):
  - Local Institution, Amsterdam
  - Local Institution, Utrecht
- Spain (5):
  - H. Univ. Vall dHebron, Barcelona
  - Fundacion Jimenez Diaz, Madrid
  - Hosp. Univ. Puerta De Hierro, Majadahonda - Madrid
  - Hospital Universitario Virgen De La Victoria, Málaga
  - Clinica Universidad de Navarra, Pamplona

REFERENCES:
- [Derived] Gutierrez M, Moreno V, Heinhuis KM, Olszanski AJ, Spreafico A, Ong M, Chu Q, Carvajal RD, Trigo J, Ochoa de Olza M, Provencio M, De Vos FY, De Braud F, Leong S, Lathers D, Wang R, Ravindran P, Feng Y, Aanur P, Melero I. OX40 Agonist BMS-986178 Alone or in Combination With Nivolumab and/or Ipilimumab in Patients With Advanced Solid Tumors. Clin Cancer Res. 2021 Jan 15;27(2):460-472. doi: 10.1158/1078-0432.CCR-20-1830. Epub 2020 Nov 4. PMID 33148673
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 165 participants were randomized and treated in Parts 1-8. 1 Participant was randomized and treated in Part 9 Cohort 1. Parts 2B, 2D, 2E, 3B, 3C, and Part 9 Cohort 2 did not enroll any participants.
Groups:
- Escalation Part 1: BMS 20 mg Q2W: Part 1A is BMS-986178 monotherapy dose escalation. Dosing of BMS-986178 20mg will begin on Day 1 of each cycle and will be administered every 2 week (q2w) for up to 12 cycles.
- Escalation Part 1: BMS 40 mg Q2W: Part 1A is BMS-986178 monotherapy dose escalation. Dosing of BMS-986178 40mg will begin on Day 1 of each cycle and will be administered every 2 week (q2w) for up to 12 cycles.
- Escalation Part 1: BMS 80 mg Q2W: Part 1A is BMS-986178 monotherapy dose escalation. Dosing of BMS-986178 80mg will begin on Day 1 of each cycle and will be administered every 2 week (q2w) for up to 12 cycles.
- Escalation Part 1: BMS 160 mg Q2W: Part 1A is BMS-986178 monotherapy dose escalation. Dosing of BMS-986178 160mg will begin on Day 1 of each cycle and will be administered every 2 week (q2w) for up to 12 cycles.
- Escalation Part 1: BMS 320 mg Q2W: Part 1A is BMS-986178 monotherapy dose escalation. Dosing of BMS-986178 320mg will begin on Day 1 of each cycle and will be administered every 2 week (q2w) for up to 12 cycles.
- Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W: Dosing of BMS-986178 20mg and Nivolumab flat dose of 240 mg will be administered every 2 weeks (q2w) starting on Day 1 of each cycle for up to 12 cycles.
- Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W: Dosing of BMS-986178 40mg and Nivolumab flat dose of 240 mg will be administered every 2 weeks (q2w) starting on Day 1 of each cycle for up to 12 cycles.
- Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W: Dosing of BMS-986178 80mg and Nivolumab flat dose of 240 mg will be administered every 2 weeks (q2w) starting on Day 1 of each cycle for up to 12 cycles.
- Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W: Dosing of BMS-986178 160mg and Nivolumab flat dose of 240 mg will be administered every 2 weeks (q2w) starting on Day 1 of each cycle for up to 12 cycles.
- Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W: Dosing of BMS-986178 320mg and Nivolumab flat dose of 240 mg will be administered every 2 weeks (q2w) starting on Day 1 of each cycle for up to 12 cycles.
- Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W: Each treatment cycle will be 3 weeks in length. BMS-986178 20mg will be administered q3w starting on Cycle 1 Day 1, up to and including 8 cycles. Ipilimumab will be administered at a dose of 1 mg/kg q3w starting on Day 1 for 4 cycles. Only BMS-986178 will be administered in the last 4 cycles.
- Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W: Each treatment cycle will be 3 weeks in length. BMS-986178 40mg will be administered q3w starting on Cycle 1 Day 1, up to and including 8 cycles. Ipilimumab will be administered at a dose of 1 mg/kg q3w starting on Day 1 for 4 cycles. Only BMS-986178 will be administered in the last 4 cycles.
- Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W: Each treatment cycle will be 3 weeks in length. BMS-986178 80mg will be administered q3w starting on Cycle 1 Day 1, up to and including 8 cycles. Ipilimumab will be administered at a dose of 1 mg/kg q3w starting on Day 1 for 4 cycles. Only BMS-986178 will be administered in the last 4 cycles.
- Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W: Each treatment cycle will be 3 weeks in length. BMS-986178 160mg will be administered q3w starting on Cycle 1 Day 1, up to and including 8 cycles. Ipilimumab will be administered at a dose of 1 mg/kg q3w starting on Day 1 for 4 cycles. Only BMS-986178 will be administered in the last 4 cycles.
- Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W: Each treatment cycle will be 3 weeks in length. BMS-986178 320mg will be administered q3w starting on Cycle 1 Day 1, up to and including 8 cycles. Ipilimumab will be administered at a dose of 1 mg/kg q3w starting on Day 1 for 4 cycles. Only BMS-986178 will be administered in the last 4 cycles.
- Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC): Participants with bladder cancer receive BMS-986178 (80 mg) and Nivolumab administered at a flat dose of 240 mg. Each treatment cycle will be 2 weeks in length and study drugs will be administered every 2 weeks starting on Day 1 of each cycle for up to 12 cycles.
- Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W: Combination arm of BMS-986178 (80 mg) with nivolumab (480 mg) to be administered every 4 weeks (q4w).
- Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W: Combination arm of BMS-986178 (80 mg) with Ipilimumab 3 mg/kg administered every 3 weeks (q3w) for 4 doses, followed by monotherapy with BMS-986178 (maintenance therapy).
- Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC): Participants with renal cell carcinoma (RCC) recieve BMS-986178 (40mg) administered at a flat dose in combination with nivolumab (240 mg) and ipilimumab (1 mg/kg) every 3 weeks (q3w) during Cycles 1 to 4, followed by maintenance therapy (Cycle 5 and beyond) in which BMS-986178 (40 mg) and nivolumab (480 mg) will be administered every 4 weeks (q4w). Study drugs will be administered accordingly starting on Day 1 of each cycle.
- Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC): Participants with renal cell carcinoma (RCC) receive BMS-986178 (40mg) administered combination with nivolumab (240 mg) and ipilimumab (1 mg/kg) every 3 weeks (q3w) during Cycles 1 to 4 followed by maintenance therapy (Cycle 5 and beyond) in which BMS-986178 and nivolumab (480 mg) will be administered every 4 weeks (q4w). Study drugs will be administered accordingly starting on Day 1 of each cycle.
- Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC): BMS-986178 will be administered at a flat dose of 40 mg (q2w) in combination with nivolumab (240 mg; q2w) and ipilimumab (1 mg/kg; q6w) for four 6-week cycles. Study drugs will be administered accordingly starting on Day 1 of each cycle. If participants continue for additional cycles, past cycle 4, all study drugs (BMS-986178/nivolumab/ipilimumab) will continue for all cycles.
- Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC): Participants with non-small cell lung cancer (NSCLC) receive BMS-986178 (40 mg) in combination with nivolumab 240 mg every 2 weeks (q2w) and ipilimumab 1 mg/kg every 6 weeks (q6w) for four, 6-week cycles. Study drugs will be administered accordingly starting on Day 1 of each cycle.
- Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W: BMS-986178 (20 mg) will be administered as a flat dose every 12 weeks (q12w) in combination with nivolumab flat dose (480 mg) every 4 weeks (q4w). Each treatment cycle will be 12 weeks in length starting on Day 1 of each cycle. There will be up to 9 cycles, to allow for 24 months of treatment. A tetanus vaccine (Tdap preferred, Td or equivalent after discussion with the medical monitor) will be administered first on Cycle 1 Day 1 prior to administration of nivolumab and BMS-986178.
- Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W: BMS-986178 (40 mg) will be administered as a flat dose every 12 weeks (q12w) in combination with nivolumab flat dose (480 mg) every 4 weeks (q4w). Each treatment cycle will be 12 weeks in length starting on Day 1 of each cycle. There will be up to 9 cycles, to allow for 24 months of treatment. A tetanus vaccine (Tdap preferred, Td or equivalent after discussion with the medical monitor) will be administered first on Cycle 1 Day 1 prior to administration of nivolumab and BMS-986178.
- Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W: BMS-986178 (80 mg) will be administered as a flat dose every 12 weeks (q12w) in combination with nivolumab flat dose (480 mg) every 4 weeks (q4w). Each treatment cycle will be 12 weeks in length starting on Day 1 of each cycle. There will be up to 9 cycles, to allow for 24 months of treatment. A tetanus vaccine (Tdap preferred, Td or equivalent after discussion with the medical monitor) will be administered first on Cycle 1 Day 1 prior to administration of nivolumab and BMS-986178.
- Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W: Nivolumab monotherapy will be administered as a flat dose of 480 mg every 4 weeks (q4w). Each treatment cycle will be 12 weeks in length and will be dosed for up to 9 cycles, 24 months of dosing. Treatment will be given on Day 1, Day 29 and 57 of each cycle. . A tetanus vaccine (Tdap preferred, Td or equivalent after discussion with the medical monitor) will be administered first on Cycle 1 Day 1 prior to administration of nivolumab monotherapy.
- Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine: Cohort 1: Cyclophosphamide 300 mg/m2 was administered 3 days prior to C1D1. DPV-001 1 mg was given on C1D1 intranodal then intradermal on C1D8, C1D15, C2D1, C2D15, C3D1, C4D1, C5D1, C6D1, C9D1 and C12D1. Nivolumab 240 mg was administered on C1D15 followed by nivolumab 480 mg was Q4W on day 1 of cycles 2-26. BMS-986178 40 mg infusion was administered on day 1 of cycles 1-6, 9, and 12. Each treatment cycle is 4 weeks and there are up to 26 cycles.
Period: Overall Study
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Started (Treated) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
Completed (Participants continuing in the study) | 3 | 4 | 4 | 3 | 3 | 4 | 8 | 10 | 7 | 8 | 3 | 6 | 5 | 6 | 5 | 15 | 10 | 2 | 5 | 1 | 4 | 8 | 2 | 1 | 1 | 1 | 0
Not Completed | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 2 | 1 | 0 | 1 | 4 | 2 | 2 | 1 | 3 | 2 | 4 | 2 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 1
Not completed — Other reasons | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Not completed — Death | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 4 | 2 | 2 | 0 | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant withdrew consent | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1 | 166
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 2 | 1 | 3 | 5 | 3 | 10 | 5 | 5 | 3 | 7 | 4 | 7 | 4 | 8 | 8 | 5 | 7 | 0 | 2 | 2 | 2 | 1 | 0 | 0 | 1 | 100
  >=65 years | 0 | 3 | 2 | 3 | 1 | 2 | 5 | 2 | 3 | 3 | 1 | 3 | 3 | 1 | 2 | 10 | 4 | 1 | 0 | 1 | 4 | 7 | 0 | 1 | 2 | 2 | 0 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 1 | 1 | 3 | 6 | 3 | 6 | 2 | 3 | 5 | 4 | 7 | 2 | 1 | 8 | 3 | 2 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 67
  Male | 3 | 3 | 1 | 3 | 3 | 4 | 2 | 9 | 2 | 6 | 1 | 5 | 3 | 1 | 4 | 17 | 4 | 3 | 5 | 1 | 4 | 9 | 2 | 1 | 1 | 2 | 0 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Not Hispanic or Latino | 3 | 4 | 4 | 3 | 2 | 6 | 6 | 5 | 3 | 3 | 2 | 7 | 4 | 4 | 5 | 6 | 5 | 3 | 0 | 1 | 4 | 3 | 1 | 2 | 1 | 1 | 1 | 89
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 6 | 5 | 5 | 2 | 3 | 1 | 4 | 1 | 12 | 7 | 3 | 6 | 0 | 2 | 6 | 1 | 0 | 1 | 1 | 0 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  White | 2 | 3 | 4 | 4 | 3 | 6 | 8 | 12 | 8 | 8 | 4 | 8 | 7 | 7 | 6 | 18 | 11 | 6 | 7 | 1 | 5 | 8 | 2 | 2 | 2 | 2 | 1 | 155
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Experiencing Dose-Limiting Toxicities (DLTs)
Description: The number of participants experiencing dose-limiting toxicities (DLTs) to assess the overall safety and tolerability of BMS-986178 administered alone or in combination with Nivolumab and/or Ipilimumab in participants with advanced solid tumors.
  DLTs are defined based on the incidence, severity, and duration of adverse events (AEs) for which no clear alternative cause is identified. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 28 days after first dose
Population: All treated participants (Parts 1-9)
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: The Number of Participants Experiencing Adverse Events (AEs)
Description: The number of participants experiencing adverse events (AEs) to assess the overall safety and tolerability of BMS-986178 administered alone or in combination with Nivolumab and/or Ipilimumab in participants with advanced solid tumors.
  An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 100 days after last dose (up to approximately 2.5 years)
Population: All treated participants (Parts 1-9)
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
Participants | 4 | 4 | 4 | 3 | 4 | 7 | 8 | 12 | 7 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 6 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1

3. Primary Outcome: The Number of Participants Experiencing Serious Adverse Events (SAEs)
Description: The number of participants experiencing serious adverse events (SAEs) to assess the overall safety and tolerability of BMS-986178 administered alone or in combination with Nivolumab and/or Ipilimumab in participants with advanced solid tumors.
  A SAE is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, and/or is an important medical event.
Time Frame: From first dose to 100 days after last dose (up to approximately 2.5 years)
Population: All treated participants (Parts 1-9)
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
Participants | 3 | 4 | 2 | 3 | 3 | 3 | 6 | 7 | 4 | 5 | 2 | 6 | 6 | 5 | 2 | 11 | 7 | 4 | 4 | 1 | 6 | 5 | 0 | 1 | 1 | 1 | 1

4. Primary Outcome: The Number of Participants Experiencing Adverse Events (AEs) Leading to Discontinuation
Description: The number of participants experiencing adverse events (AEs) leading to discontinuation of study drug to assess the overall safety and tolerability of BMS-986178 administered alone or in combination with Nivolumab and/or Ipilimumab in participants with advanced solid tumors. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 100 days after last dose (up to approximately 2.5 years)
Population: All treated participants (Parts 1-9)
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: The Number of Participant Deaths
Description: The number of deaths in each arm to assess the overall safety and tolerability of BMS-986178 administered alone or in combination with Nivolumab and/or Ipilimumab in participants with advanced solid tumors.
Time Frame: From first dose to study completion (up to approximately 4 years 5 months)
Population: All treated participants (Parts 1-9)
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
Participants | 4 | 4 | 3 | 4 | 4 | 3 | 7 | 11 | 6 | 6 | 4 | 9 | 7 | 8 | 2 | 16 | 11 | 3 | 3 | 0 | 5 | 4 | 2 | 2 | 1 | 1 | 1

6. Primary Outcome: The Number of Participants With Clinical Laboratory Test Abnormalities (Hematology)
Description: The number of participants with clinical laboratory test abnormalities to assess the overall safety and tolerability of BMS-986178 administered alone or in combination with Nivolumab and/or Ipilimumab in participants with advanced solid tumors.
  Results will be categorized according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.
  Grade 1 = Mild Grade 2 = Moderate Grade 3 = Severe Grade 4 = Life Threatening Grade 5 = Death Related to AE Baseline is defined as the last non-missing measurement prior to the first dosing date and time
Time Frame: From baseline to 100 days after last dose (up to approximately 2.5 years)
Population: All treated participants with on-treatment laboratory results and CTC grade criteria available (Parts 1-9)
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
Participants
  HEMOGLOBIN GRADE 1 | 2 | 0 | 4 | 1 | 2 | 1 | 4 | 3 | 3 | 6 | 3 | 4 | 2 | 5 | 1 | 9 | 4 | 1 | 3 | 1 | 2 | 7 | 1 | 1 | 1 | 1 | 1
  HEMOGLOBIN GRADE 2 | 1 | 2 | 0 | 2 | 1 | 4 | 2 | 5 | 2 | 0 | 1 | 6 | 3 | 1 | 4 | 6 | 5 | 2 | 2 | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 0
  HEMOGLOBIN GRADE 3 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 2 | 1 | 3 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
  PLATELET COUNT GRADE 1: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  PLATELET COUNT GRADE 1 | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 2 | 4 | 3 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
  PLATELET COUNT GRADE 2: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 00
  PLATELET COUNT GRADE 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  PLATELET COUNT GRADE 3: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  PLATELET COUNT GRADE 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LEUKOCYTES GRADE 1: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  LEUKOCYTES GRADE 1 | 1 | 1 | 2 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 1 | 1 | 3 | 2 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
  LEUKOCYTES GRADE 2: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  LEUKOCYTES GRADE 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
  LEUKOCYTES GRADE 3: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  LEUKOCYTES GRADE 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LEUKOCYTES GRADE 4: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  LEUKOCYTES GRADE 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ABSOLUTE NEUTROPHIL COUNT DRV. GRADE 1: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  ABSOLUTE NEUTROPHIL COUNT DRV. GRADE 1 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  ABSOLUTE NEUTROPHIL COUNT DRV. GRADE 2: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  ABSOLUTE NEUTROPHIL COUNT DRV. GRADE 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ABSOLUTE NEUTROPHIL COUNT DRV. GRADE 3: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  ABSOLUTE NEUTROPHIL COUNT DRV. GRADE 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  ABSOLUTE NEUTROPHIL COUNT DRV. GRADE 4: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  ABSOLUTE NEUTROPHIL COUNT DRV. GRADE 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: The Number of Participants With Clinical Laboratory Test Abnormalities (LIVER AND KIDNEY FUNCTION)
Description: as for outcome 6
Time Frame: From baseline to 100 days after last dose (up to approximately 2.5 years)
Population: All treated participants with on-treatment laboratory results and CTC grade criteria available (Parts 1-9)
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
Participants
  ALKALINE PHOSPHATASE GRADE 1 | 2 | 2 | 2 | 1 | 3 | 5 | 2 | 5 | 6 | 4 | 2 | 3 | 3 | 4 | 0 | 7 | 6 | 2 | 1 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 1
  ALKALINE PHOSPHATASE GRADE 2 | 1 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 3 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 1
  ALKALINE PHOSPHATASE GRADE 3 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  ASPARTATE AMINOTRANSFERASE GRADE 1 | 2 | 3 | 1 | 1 | 1 | 3 | 4 | 2 | 1 | 2 | 0 | 4 | 2 | 2 | 2 | 10 | 5 | 4 | 3 | 0 | 5 | 2 | 0 | 1 | 1 | 0 | 1
  ASPARTATE AMINOTRANSFERASE GRADE 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  ASPARTATE AMINOTRANSFERASE GRADE 3 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ASPARTATE AMINOTRANSFERASE GRADE 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALANINE AMINOTRANSFERASE GRADE 1 | 1 | 3 | 2 | 2 | 0 | 2 | 4 | 1 | 2 | 0 | 1 | 4 | 1 | 1 | 2 | 7 | 4 | 3 | 1 | 0 | 3 | 3 | 0 | 1 | 0 | 0 | 1
  ALANINE AMINOTRANSFERASE GRADE 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALANINE AMINOTRANSFERASE GRADE 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALANINE AMINOTRANSFERASE GRADE 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BILIRUBIN, TOTAL GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BILIRUBIN, TOTAL GRADE 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  BILIRUBIN, TOTAL GRADE 3 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BILIRUBIN, TOTAL GRADE 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CREATININE GRADE 1 | 2 | 1 | 2 | 1 | 0 | 0 | 3 | 6 | 1 | 1 | 0 | 1 | 1 | 3 | 2 | 7 | 0 | 1 | 2 | 1 | 2 | 3 | 1 | 1 | 1 | 1 | 0
  CREATININE GRADE 2: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  CREATININE GRADE 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  CREATININE GRADE 3: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  CREATININE GRADE 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: The Number of Participants With Clinical Laboratory Test Abnormalities (OTHER CHEMISTRY TESTING )
Description: as for outcome 6
Time Frame: From baseline to 100 days after last dose (up to approximately 2.5 years)
Population: All treated participants with on-treatment laboratory results and CTC grade criteria available (Parts 1-9)
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
Participants
  SODIUM, SERUM GRADE 1 | 4 | 3 | 2 | 2 | 1 | 2 | 6 | 5 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 4 | 3 | 1 | 0 | 0 | 4 | 1 | 0 | 1 | 0 | 1 | 1
  SODIUM, SERUM GRADE 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SODIUM, SERUM GRADE 3 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  POTASSIUM, SERUM GRADE 1: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  POTASSIUM, SERUM GRADE 1 | 0 | 3 | 0 | 2 | 0 | 1 | 4 | 3 | 2 | 2 | 0 | 2 | 3 | 2 | 2 | 8 | 3 | 0 | 1 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0
  POTASSIUM, SERUM GRADE 2: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  POTASSIUM, SERUM GRADE 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  POTASSIUM, SERUM GRADE 3: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  POTASSIUM, SERUM GRADE 3 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  POTASSIUM, SERUM GRADE 4: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  POTASSIUM, SERUM GRADE 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CALCIUM, TOTAL GRADE 1: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  CALCIUM, TOTAL GRADE 1 | 0 | 3 | 1 | 1 | 1 | 3 | 5 | 4 | 2 | 4 | 2 | 4 | 3 | 0 | 2 | 9 | 4 | 1 | 4 | 0 | 1 | 5 | 1 | 0 | 0 | 0 | 0
  CALCIUM, TOTAL GRADE 2: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  CALCIUM, TOTAL GRADE 2 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  CALCIUM, TOTAL GRADE 3: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  CALCIUM, TOTAL GRADE 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MAGNESIUM, SERUM GRADE 1: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  MAGNESIUM, SERUM GRADE 1 | 1 | 1 | 0 | 2 | 2 | 0 | 1 | 3 | 4 | 1 | 2 | 4 | 0 | 0 | 2 | 6 | 2 | 2 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 2 | 0
  MAGNESIUM, SERUM GRADE 2: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  MAGNESIUM, SERUM GRADE 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MAGNESIUM, SERUM GRADE 3: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  MAGNESIUM, SERUM GRADE 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  GLUCOSE, FASTING SERUM GRADE 1: number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 5 | 7 | 6 | 3 | 2 | 3 | 7 | 6 | 5 | 3 | 3 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
  GLUCOSE, FASTING SERUM GRADE 1 | 1 | 3 | 0 | 3 | 1 | 4 | 4 | 2 | 2 | 0 | 2 | 6 | 5 | 2 | 2 | 2 |  |  | 0 |  | 0 | 0 |  |  |  |  | 0
  GLUCOSE, FASTING SERUM GRADE 2: number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 5 | 7 | 6 | 3 | 2 | 3 | 7 | 6 | 5 | 3 | 3 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
  GLUCOSE, FASTING SERUM GRADE 2 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 |  |  | 0 |  | 1 | 0 |  |  |  |  | 0
  GLUCOSE, FASTING SERUM GRADE 3: number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 5 | 7 | 6 | 3 | 2 | 3 | 7 | 6 | 5 | 3 | 3 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
  GLUCOSE, FASTING SERUM GRADE 3 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  | 0 |  | 0 | 0 |  |  |  |  | 0
  ALBUMIN GRADE 1 | 2 | 2 | 1 | 2 | 1 | 2 | 0 | 4 | 1 | 3 | 1 | 2 | 5 | 2 | 1 | 3 | 4 | 2 | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 1 | 0
  ALBUMIN GRADE 2 | 1 | 2 | 2 | 1 | 1 | 3 | 5 | 3 | 3 | 0 | 2 | 4 | 1 | 2 | 3 | 5 | 2 | 2 | 2 | 1 | 3 | 4 | 0 | 0 | 0 | 1 | 1
  ALBUMIN GRADE 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  AMYLASE, TOTAL GRADE 1: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  AMYLASE, TOTAL GRADE 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  AMYLASE, TOTAL GRADE 2: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  AMYLASE, TOTAL GRADE 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  AMYLASE, TOTAL GRADE 3: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  AMYLASE, TOTAL GRADE 3 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AMYLASE, TOTAL GRADE 4: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  AMYLASE, TOTAL GRADE 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  LIPASE, TOTAL GRADE 1: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  LIPASE, TOTAL GRADE 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0
  LIPASE, TOTAL GRADE 2: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  LIPASE, TOTAL GRADE 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LIPASE, TOTAL GRADE 3: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  LIPASE, TOTAL GRADE 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
  LIPASE, TOTAL GRADE 4: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 0
  LIPASE, TOTAL GRADE 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

9. Secondary Outcome: Objective Response Rate (ORR)
Description: The total number of participants whose best overall response (BOR) is either a complete response (CR) or partial response (PR) based on assessment of tumor response using RECIST v1.1.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions:
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions.
  Overall Response (OR) = CR + PR Baseline is defined as the last non-missing measurement prior to the first dosing date and time.
Time Frame: From baseline up to approximately 2.5 years
Population: Response Evaluable Participants (Parts 1-9)
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 9 | 8 | 8 | 5 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | NA — BOR was not evaluable for the patient due to death prior to any tumor assessment

10. Secondary Outcome: Duration of Response (DOR)
Description: The time between the date of first response and the subsequent date of disease progression or death (death after re-treatment will not be considered), whichever occurs first in participants with a best overall response (BOR) of complete response (CR) or partial response (PR).
  Best overall response (BOR) is assessed per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions:
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions.
  Baseline is defined as the last non-missing measurement prior to the first dosing date and time.
  Due to high percentage of censored response, median estimate may be misleading
Time Frame: From baseline up to approximately 2.5 years
Population: The number of responders within each tumor type was not sufficient for analysis. (Parts 1-8)
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weeks |  |  |  |  |  |  | NA [NA to NA] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | 17.14 [NA to NA] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [NA to NA] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. | NA [NA to NA] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. |  |  |  |  |  | NA [NA to NA] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. |  |  | 64.14 [NA to NA] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. |  |  | NA [NA to NA] — KM methodology requires having more than 50% of events to estimate the median and/or upper/lower limits. |  |  |  |

11. Secondary Outcome: Progression Free Survival (PFS) Rate at 24 Weeks
Description: The percentage of treated participants remaining progression free and surviving at 24 weeks since the first dosing date.
Time Frame: 24 weeks after first dose
Population: All treated Participants (Parts 1-8)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2
Percentage of participants | 0.0 [NA to NA] — The estimate (or confidence of estimate) is N.A because no observations were available for calculation of estimate (or confidence of estimate).) | 0.0 [NA to NA] — The estimate (or confidence of estimate) is N.A because no observations were available for calculation of estimate (or confidence of estimate). | 0.0 [NA to NA] — The estimate (or confidence of estimate) is N.A because no observations were available for calculation of estimate (or confidence of estimate). | 25.0 [0.9 to 66.5] | 25.0 [0.9 to 66.5] | 17.9 [0.8 to 53.8] | 42.9 [9.8 to 73.4] | 16.7 [2.7 to 41.3] | 28.6 [4.1 to 61.2] | 37.5 [8.7 to 67.4] | 0.0 [NA to NA] — The estimate (or confidence of estimate) is N.A because no observations were available for calculation of estimate (or confidence of estimate). | 11.1 [0.6 to 38.8] | 0.0 [NA to NA] — The estimate (or confidence of estimate) is N.A because no observations were available for calculation of estimate (or confidence of estimate). | 0.0 [NA to NA] — The estimate (or confidence of estimate) is N.A because no observations were available for calculation of estimate (or confidence of estimate). | 40.0 [5.2 to 75.3] | 22.2 [6.9 to 42.9] | 9.2 [0.5 to 33.5] | 0.0 [NA to NA] — The estimate (or confidence of estimate) is N.A because no observations were available for calculation of estimate (or confidence of estimate). | 28.6 [4.1 to 61.2] | NA [NA to NA] — The estimate (or confidence of estimate) is N.A because no observations were available for calculation of estimate (or confidence of estimate). | 0.0 [NA to NA] — The estimate (or confidence of estimate) is N.A because no observations were available for calculation of estimate (or confidence of estimate). | 33.3 [7.8 to 62.3] | 0.0 [NA to NA] — The estimate (or confidence of estimate) is N.A because no observations were available for calculation of estimate (or confidence of estimate). | 0.0 [NA to NA] — The estimate (or confidence of estimate) is N.A because no observations were available for calculation of estimate (or confidence of estimate). | 0.0 [NA to NA] — The estimate (or confidence of estimate) is N.A because no observations were available for calculation of estimate (or confidence of estimate). | 50.0 [0.6 to 91.0]

12. Secondary Outcome: Cmax: Maximum Observed Serum Concentration
Description: The maximum observed serum concentration was measured after dosing to assess the pharmacokinetics of BMS-986178 administered alone or in combination with Nivolumab and/or Ipilimumab.
  Note: The geometric CV was not calculated. Arithmetic % CV is reported instead.
Time Frame: Cycle 1-9 timepoints can include (Pre-dose, 0.30, 4, 24, 72, 168, 336, 696 hours post dose)
Population: Pharmacokinetic participants: All participants with available serum time-concentration data from subjects who received any BMS-986178 or Nivolumab or Ipilimumab. (Parts 1-9)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: NG/ML
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
NG/ML
  CYCLE 1 DAY 1: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 9 | 7 | 8 | 6 | 18 | 9 | 6 | 6 | 0 | 5 | 8 | 1 | 1 | 0 | 0 | 0
  CYCLE 1 DAY 1 | 4964 (11) | 11245 (34) | 19254 (18) | 36143 (14) | 68774 (20) | 9424 (133) | 11699 (13) | 19547 (39) | 39182 (37) | 76445 (22) | 7860 (35) | 9345 (20) | 17979 (31) | 55790 (107) | 65472 (27) | 17586 (25) | 19012 (22) | 21399 (12) | 11139 (19) |  | 14267 (37) | 15424 (173) | 3270 (NA) — No measure of variation/dispersion for a single data value | 11300 (NA) — No measure of variation/dispersion for a single data value |  |  |
  CYCLE 4 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 3 | 2 | 0 | 0 | 1 | 3 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0
  CYCLE 4 DAY 1 |  |  |  |  |  |  |  |  |  |  | 8960 (NA) — No measure of variation/dispersion for a single data value | 10273 (12) | 20900 (NA) — No measure of variation/dispersion for a single data value | 69922 (36) | 117839 (15) |  |  | 31800 (NA) — No measure of variation/dispersion for a single data value | 11261 (21) |  |  | 14143 (47) |  |  |  |  |
  CYCLE 5 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 5 DAY 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 16912 (36) |  |  |  |  |  |  |  |  |  |
  CYCLE 9 DAY 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 9 DAY 1 |  |  | 23200 (NA) — No measure of variation/dispersion for a single data value | 61500 (NA) — No measure of variation/dispersion for a single data value |  |  | 17392 (19) | 23097 (66) | 72991 (12) | 207853 (33) |  |  |  |  |  | 30922 (30) |  |  |  |  |  |  |  |  |  |  |

13. Secondary Outcome: Tmax: Time of Maximum Observed Serum Concentration
Description: The time of maximum observed serum concentration was measured after dosing to assess the pharmacokinetics of BMS-986178 administered alone or in combination with Nivolumab and/or Ipilimumab
Time Frame: Cycle 1-9 timepoints can include (Pre-dose, 0.30, 4, 24, 72, 168, 336, 696 hours post dose)
Population: as for outcome 12
Measure: Median (Full Range); unit: Hours
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
Hours
  CYCLE 1 DAY 1: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 9 | 7 | 8 | 6 | 18 | 9 | 6 | 6 | 0 | 5 | 8 | 1 | 1 | 0 | 0 | 0
  CYCLE 1 DAY 1 | 0.675 [0.467 to 4.52] | 0.575 [0.467 to 0.933] | 4.58 [0.500 to 24.0] | 2.30 [0.567 to 4.02] | 0.558 [0.467 to 4.08] | 0.467 [0.467 to 4.00] | 2.34 [0.467 to 4.08] | 0.517 [0.467 to 4.50] | 0.650 [0.517 to 4.10] | 0.792 [0.450 to 4.50] | 0.667 [0.633 to 4.08] | 4.00 [0.467 to 4.13] | 4.00 [0.467 to 4.43] | 2.55 [0.467 to 24.1] | 4.13 [0.467 to 4.62] | 4.09 [0.467 to 4.82] | 0.550 [0.500 to 24.0] | 2.30 [0.467 to 4.55] | 0.583 [0.467 to 4.08] |  | 4.00 [0.517 to 23.0] | 0.475 [0.467 to 4.75] | 0.533 [0.533 to 0.533] | 4.83 [4.83 to 4.83] |  |  |
  CYCLE 4 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 3 | 2 | 0 | 0 | 1 | 3 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0
  CYCLE 4 DAY 1 |  |  |  |  |  |  |  |  |  |  | 0.583 [0.583 to 0.583] | 4.00 [0.617 to 24.0] | 0.583 [0.583 to 0.583] | 4.00 [0.467 to 24.9] | 2.58 [0.467 to 4.68] |  |  | 4.03 [4.03 to 4.03] | 0.517 [0.500 to 0.583] |  |  | 0.467 [0.000 to 4.00] |  |  |  |  |
  CYCLE 5 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 5 DAY 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0.550 [0.517 to 0.583] |  |  |  |  |  |  |  |  |  |
  CYCLE 9 DAY 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 9 DAY 1 |  |  | 0.467 [0.467 to 0.467] | 22.7 [22.7 to 22.7] |  |  | 0.567 [0.467 to 4.00] | 4.47 [4.02 to 4.50] | 2.38 [0.633 to 4.12] | 4.05 [3.98 to 23.9] |  |  |  |  |  | 3.94 [0.500 to 4.03] |  |  |  |  |  |  |  |  |  |  |

14. Secondary Outcome: AUC(0-t): Area Under the Serum Concentration-time Curve From Time 0 to Time t
Description: The area under the serum concentration-time curve from time 0 to time t was measured after dosing to assess the pharmacokinetics of BMS-986178 administered alone or in combination with Nivolumab and/or Ipilimumab.
  Note: The geometric CV was not calculated. Arithmetic % CV is reported instead.
Time Frame: Cycle 1-9 timepoints can include (Pre-dose, 0.30, 4, 24, 72, 168, 336, 696 hours post dose)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: H*NG/ML
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
H*NG/ML
  CYCLE 1 DAY 1: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 9 | 7 | 8 | 6 | 18 | 9 | 6 | 6 | 0 | 5 | 8 | 1 | 1 | 0 | 0 | 0
  CYCLE 1 DAY 1 | 577541 (31) | 1678196 (23) | 1825502 (61) | 5024906 (32) | 9981469 (9) | 609426 (62) | 1495494 (27) | 2324225 (24) | 5458640 (47) | 8694104 (46) | 1047354 (49) | 1197507 (43) | 2774058 (56) | 7257441 (34) | 10580541 (41) | 2351794 (29) | 2000522 (43) | 3216650 (21) | 1251698 (49) |  | 1653102 (22) | 864500 (57) | 390424 (NA) — No measure of variation/dispersion for a single data value | 2399055 (NA) — No measure of variation/dispersion for a single data value |  |  |
  CYCLE 4 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 3 | 2 | 0 | 0 | 1 | 3 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0
  CYCLE 4 DAY 1 |  |  |  |  |  |  |  |  |  |  | 773957 (NA) — No measure of variation/dispersion for a single data value | 2210404 (21) | 2400433 (NA) — No measure of variation/dispersion for a single data value | 10729551 (38) | 23851864 (14) |  |  | 2699238 (NA) — No measure of variation/dispersion for a single data value | 1837861 (10) |  |  | 504998 (91) |  |  |  |  |
  CYCLE 5 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 5 DAY 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 2520673 (50) |  |  |  |  |  |  |  |  |  |
  CYCLE 9 DAY 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 9 DAY 1 |  |  | 3952990 (NA) — No measure of variation/dispersion for a single data value | 13024914 (NA) — No measure of variation/dispersion for a single data value |  |  | 2971409 (53) | 1247687 (118) | 16483279 (37) | 28499982 (78) |  |  |  |  |  | 4537054 (42) |  |  |  |  |  |  |  |  |  |  |

15. Secondary Outcome: AUC(TAU): Area Under the Serum Concentration-time Curve in 1 Dosing Interval
Description: The area under the serum concentration-time curve in 1 dosing interval was measured after dosing to assess the pharmacokinetics of BMS-986178 administered alone or in combination with Nivolumab and/or Ipilimumab.
  Note: The geometric CV was not calculated. Arithmetic % CV is reported instead.
Time Frame: Cycle 1-9 timepoints can include (Pre-dose, 0.30, 4, 24, 72, 168, 336, 696 hours post dose)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: H*NG/ML
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
H*NG/ML
  CYCLE 1 DAY 1: number analyzed (Participants) | 4 | 4 | 3 | 3 | 4 | 6 | 8 | 11 | 8 | 6 | 3 | 6 | 6 | 8 | 5 | 15 | 6 | 6 | 5 | 0 | 3 | 6 | 1 | 1 | 0 | 0 | 0
  CYCLE 1 DAY 1 | 577541 (31) | 1599886 (29) | 3142196 (21) | 5854143 (19) | 9981469 (9) | 663257 (60) | 1515139 (24) | 2551115 (24) | 5458640 (47) | 11483961 (26) | 1383126 (28) | 1521223 (31) | 3133192 (49) | 7464248 (32) | 11966698 (34) | 2602049 (23) | 2734577 (31) | 3500606 (28) | 1568004 (33) |  | 1705864 (10) | 1410042 (23) | 447709 (NA) — No measure of variation/dispersion for a single data value | 2812249 (NA) — No measure of variation/dispersion for a single data value |  |  |
  CYCLE 4 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
  CYCLE 4 DAY 1 |  |  |  |  |  |  |  |  |  |  |  | 2210404 (21) |  | 12666237 (39) | 27936423 (8) |  |  |  | 1837861 (10) |  |  | 3590883 (12) |  |  |  |  |
  CYCLE 5 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 5 DAY 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 3335668 (56) |  |  |  |  |  |  |  |  |  |
  CYCLE 9 DAY 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 9 DAY 1 |  |  | 3952990 (NA) — No measure of variation/dispersion for a single data value | 13024914 (NA) — No measure of variation/dispersion for a single data value |  |  | 3345948 (40) | 3307867 (83) | 16483279 (37) | 50254284 (42) |  |  |  |  |  | 6176469 (17) |  |  |  |  |  |  |  |  |  |  |

16. Secondary Outcome: Ctau: Observed Serum Concentration at the End of a Dosing Interval When Intensive Samples Are Collected
Description: The observed serum concentration at the end of a dosing interval when intensive samples are collected was measured after dosing to assess the pharmacokinetics of BMS-986178 administered alone or in combination with Nivolumab and/or Ipilimumab.
  Note: The geometric CV was not calculated. Arithmetic % CV is reported instead.
Time Frame: Cycle 1-9 timepoints can include (Pre-dose, 0.30, 4, 24, 72, 168, 336, 696 hours post dose)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: NG/ML
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
NG/ML
  CYCLE 1 DAY 1: number analyzed (Participants) | 4 | 4 | 3 | 3 | 4 | 6 | 8 | 11 | 8 | 6 | 3 | 6 | 6 | 8 | 5 | 15 | 6 | 6 | 5 | 0 | 3 | 6 | 1 | 1 | 0 | 0 | 0
  CYCLE 1 DAY 1 | 657 (62) | 2577 (30) | 5354 (31) | 10852 (44) | 16514 (4) | 756 (108) | 1904 (37) | 3598 (37) | 10413 (51) | 18596 (41) | 885 (56) | 604 (67) | 2335 (87) | 3059 (93) | 7739 (72) | 3928 (33) | 544 (76) | 1725 (76) | 790 (88) |  | 1535 (35) | 1533 (54) | 0.004 (NA) — No measure of variation/dispersion for a single data value | 42.9 (NA) — No measure of variation/dispersion for a single data value |  |  |
  CYCLE 4 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
  CYCLE 4 DAY 1 |  |  |  |  |  |  |  |  |  |  |  | 2527 (68) |  | 7729 (49) | 32982 (33) |  |  |  | 1262 (10) |  |  | 6906 (20) |  |  |  |  |
  CYCLE 5 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 5 DAY 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1412 (78) |  |  |  |  |  |  |  |  |  |
  CYCLE 9 DAY 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 9 DAY 1 |  |  | 6470 (NA) — No measure of variation/dispersion for a single data value | 33600 (NA) — No measure of variation/dispersion for a single data value |  |  | 5510 (68) | 5686 (78) | 34303 (25) | 131520 (70) |  |  |  |  |  | 13400 (26) |  |  |  |  |  |  |  |  |  |  |

17. Secondary Outcome: CLT: Total Body Clearance
Description: The total body clearance was measured after dosing to assess the pharmacokinetics of BMS-986178 administered alone or in combination with Nivolumab and/or Ipilimumab.
  Note: The geometric CV was not calculated. Arithmetic % CV is reported instead.
Time Frame: Cycle 1-9 timepoints can include (Pre-dose, 0.30, 4, 24, 72, 168, 336, 696 hours post dose)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/H
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
L/H
  CYCLE 4 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
  CYCLE 4 DAY 1 |  |  |  |  |  |  |  |  |  |  |  | 0.018 (24) |  | 0.013 (44) | 0.011 (8) |  |  |  | 0.022 (10) |  |  | 0.011 (13) |  |  |  |  |
  CYCLE 5 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 5 DAY 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0.024 (56) |  |  |  |  |  |  |  |  |  |
  CYCLE 9 DAY 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 9 DAY 1 |  |  | 0.020 (NA) — No measure of variation/dispersion for a single data value | 0.012 (NA) — No measure of variation/dispersion for a single data value |  |  | 0.012 (38) | 0.024 (83) | 0.010 (37) | 0.006 (42) |  |  |  |  |  | 0.013 (19) |  |  |  |  |  |  |  |  |  |  |

18. Secondary Outcome: Css-avg: Average Concentration Over a Dosing Interval (AUC(TAU)/Tau)
Description: The average concentration over a dosing interval (AUC(TAU)/tau) was measured after dosing to assess the pharmacokinetics of BMS-986178 administered alone or in combination with Nivolumab and/or Ipilimumab.
  Note: The geometric CV was not calculated. Arithmetic % CV is reported instead.
Time Frame: Cycle 1-9 timepoints can include (Pre-dose, 0.30, 4, 24, 72, 168, 336, 696 hours post dose)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: NG/ML
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
NG/ML
  CYCLE 4 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
  CYCLE 4 DAY 1 |  |  |  |  |  |  |  |  |  |  |  | 4379 (21) |  | 25131 (39) | 55386 (8) |  |  |  | 3715 (10) |  |  | 10739 (12) |  |  |  |  |
  CYCLE 5 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 5 DAY 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 4964 (56) |  |  |  |  |  |  |  |  |  |
  CYCLE 9 DAY 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 9 DAY 1 |  |  | 11826 (NA) — No measure of variation/dispersion for a single data value | 45155 (NA) — No measure of variation/dispersion for a single data value |  |  | 9746 (42) | 9903 (83) | 45878 (27) | 148579 (42) |  |  |  |  |  | 19538 (19) |  |  |  |  |  |  |  |  |  |  |

19. Secondary Outcome: AI: Accumulation Index. Ratio of an Exposure Measure at Steady State (Cmax)
Description: The ratio of an exposure measure at steady state to that after the first dose was measured after dosing to assess the pharmacokinetics of BMS-986178 administered alone or in combination with Nivolumab and/or Ipilimumab.
  Note: The geometric CV was not calculated. Arithmetic % CV is reported instead.
Time Frame: Cycle 1-9 timepoints can include (Pre-dose, 0.30, 4, 24, 72, 168, 336, 696 hours post dose)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: NG/ML
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
NG/ML
  CYCLE 4 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 3 | 2 | 0 | 0 | 1 | 3 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0
  CYCLE 4 DAY 1 |  |  |  |  |  |  |  |  |  |  | 0.793 (NA) — No measure of variation/dispersion for a single data value | 1.05 (21) | 1.67 (NA) — No measure of variation/dispersion for a single data value | 1.40 (18) | 1.52 (18) |  |  | 1.32 (NA) — No measure of variation/dispersion for a single data value | 1.03 (15) |  |  | 1.21 (43) |  |  |  |  |
  CYCLE 5 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 5 DAY 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1.02 (5) |  |  |  |  |  |  |  |  |  |
  CYCLE 9 DAY 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 9 DAY 1 |  |  | 1.45 (NA) — No measure of variation/dispersion for a single data value | 1.89 (NA) — No measure of variation/dispersion for a single data value |  |  | 1.40 (22) | 1.29 (66) | 1.83 (14) | 2.56 (29) |  |  |  |  |  | 1.66 (32) |  |  |  |  |  |  |  |  |  |  |

20. Secondary Outcome: AI: Accumulation Index. Ratio of an Exposure Measure at Steady State (AUC)
Description: as for outcome 19
Time Frame: Cycle 1-9 timepoints can include (Pre-dose, 0.30, 4, 24, 72, 168, 336, 696 hours post dose)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: H*NG/ML
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
H*NG/ML
  CYCLE 4 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 2 | 0 | 0 | 1 | 3 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
  CYCLE 4 DAY 1 |  |  |  |  |  |  |  |  |  |  |  | 1.28 (7) |  | 1.56 (19) | 1.77 (27) |  |  | 0.000 (NA) — No measure of variation/dispersion for a single data value | 1.37 (12) |  |  | 2.13 (116) |  |  |  |  |
  CYCLE 5 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 5 DAY 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1.21 (34) |  |  |  |  |  |  |  |  |  |
  CYCLE 9 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 9 DAY 1 |  |  |  | 2.21 (NA) — No measure of variation/dispersion for a single data value |  |  | 1.85 (24) | 0.748 (141) | 2.78 (34) | 4.40 (87) |  |  |  |  |  | 2.32 (9) |  |  |  |  |  |  |  |  |  |  |

21. Secondary Outcome: AI: Accumulation Index. Ratio of an Exposure Measure at Steady State (Ctau)
Description: as for outcome 19
Time Frame: Cycle 1-9 timepoints can include (Pre-dose, 0.30, 4, 24, 72, 168, 336, 696 hours post dose)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: NG/ML
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
NG/ML
  CYCLE 4 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 2 | 0 | 0 | 1 | 3 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
  CYCLE 4 DAY 1 |  |  |  |  |  |  |  |  |  |  |  | 1.90 (73) |  | 1.22 (16) | 1.89 (29) |  |  | 0.000 (NA) — No measure of variation/dispersion for a single data value | 2.47 (57) |  |  | 2.72 (116) |  |  |  |  |
  CYCLE 5 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 5 DAY 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1.05 (48) |  |  |  |  |  |  |  |  |  |
  CYCLE 9 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 9 DAY 1 |  |  |  | 2.33 (NA) — No measure of variation/dispersion for a single data value |  |  | 2.40 (36) | 1.22 (141) | 2.61 (11) | 7.55 (87) |  |  |  |  |  | 3.49 (11) |  |  |  |  |  |  |  |  |  |  |

22. Secondary Outcome: T-HALFeff: Effective Elimination Half-life That Explains the Degree of Accumulation Observed for a Specific Exposure Measure (Exposure Measure Includes AUC(TAU), Cmax)
Description: The effective elimination half-life that explains the degree of accumulation observed for a specific exposure measure was measured after dosing to assess the pharmacokinetics of BMS-986178 administered alone or in combination with Nivolumab and/or Ipilimumab
Time Frame: Cycle 1-9 timepoints can include (Pre-dose, 0.30, 4, 24, 72, 168, 336, 696 hours post dose)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Hr
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
Hr
  CYCLE 4 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 2 | 0 | 0 | 1 | 3 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0
  CYCLE 4 DAY 1 |  |  |  |  |  |  |  |  |  |  |  | 229 (40) |  | 345 (111) | 429 (182) |  |  | 0.000 (NA) — No measure of variation/dispersion for a single data value | 261 (58) |  |  | 146 (200) |  |  |  |  |
  CYCLE 5 DAY 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 5 DAY 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 447 (NA) — No measure of variation/dispersion for a single data value |  |  |  |  |  |  |  |  |  |
  CYCLE 9 DAY 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 9 DAY 1 |  |  | 0.000 (NA) — No measure of variation/dispersion for a single data value | 331 (NA) — No measure of variation/dispersion for a single data value |  |  | 315 (119) | 0.000 (0.000) | 593 (308) | 607 (527) |  |  |  |  |  | 312 (180) |  |  |  |  |  |  |  |  |  |  |

23. Secondary Outcome: Ctrough: Trough Observed Plasma Concentration
Description: Trough observed plasma concentration (this includes predose concentrations and Ctau concentrations) was measured after dosing to assess the pharmacokinetics of BMS-986178 administered alone or in combination with Nivolumab and/or Ipilimumab.
  Note: The geometric CV was not calculated. Arithmetic % CV is reported instead.
Time Frame: Cycle 1-17 timepoints can include (Pre-dose, 336, 504, 672 hours post dose)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 7 | 8 | 12 | 8 | 8 | 4 | 10 | 7 | 8 | 6 | 18 | 12 | 6 | 7 | 1 | 6 | 9 | 2 | 2 | 2 | 2 | 1
ng/mL
  CYCLE 1 DAY 15 336 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 0 | 0 | 0 | 0 | 0
  CYCLE 1 DAY 15 336 h |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1535 (34.9) | 1912 (45.2) |  |  |  |  |
  CYCLE 1 DAY 29 0 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 7 | 0 | 0 | 0 | 0 | 0
  CYCLE 1 DAY 29 0 h |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1354 (65.0) | 1108 (72.9) |  |  |  |  |
  CYCLE 2 DAY 1 0 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 7 | 0 | 0 | 0 | 0 | 0
  CYCLE 2 DAY 1 0 h |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1391 (63.3) | 1107 (84.5) |  |  |  |  |
  CYCLE 2 DAY 1 336 h: number analyzed (Participants) | 4 | 4 | 3 | 3 | 4 | 5 | 7 | 9 | 8 | 6 | 0 | 0 | 0 | 0 | 0 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 2 DAY 1 336 h | 657 (62.2) | 2372 (38.9) | 5354 (31.0) | 10852 (44.3) | 16514 (4.14) | 561 (119) | 1995 (35.1) | 4006 (31.0) | 10413 (51.3) | 18596 (41.4) |  |  |  |  |  | 4070 (30.7) |  |  |  |  |  |  |  |  |  |  |
  CYCLE 2 DAY 1 504 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 7 | 5 | 7 | 5 | 0 | 0 | 3 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 2 DAY 1 504 h |  |  |  |  |  |  |  |  |  |  | 456 (85.5) | 591 (76.7) | 2401 (86.0) | 1921 (103) | 7739 (72.3) |  |  | 2166 (33.7) | 745 (90.9) | 1030 (NA) — No measure of variation/dispersion for a single data value |  |  |  |  |  |  |
  CYCLE 2 DAY 1 672 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 2 DAY 1 672 h |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 676 (105) |  |  |  |  |  |  |  |  |  |
  CYCLE 3 DAY 1 0 h: number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 4 | 6 | 8 | 7 | 7 | 3 | 4 | 4 | 4 | 3 | 14 | 4 | 1 | 4 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0
  CYCLE 3 DAY 1 0 h | 1290 (43.3) | 4244 (36.2) | 5903 (45.5) | 16974 (28.9) | 21571 (15.9) | 614 (122) | 1825 (70.1) | 4498 (45.4) | 16379 (43.6) | 28282 (43.2) | 323 (101) | 2049 (40.1) | 4894 (60.7) | 2766 (99.8) | 20410 (42.5) | 5055 (46.8) | 1480 (81.5) | 62.5 (NA) — No measure of variation/dispersion for a single data value | 689 (123) |  |  | 2469 (64.6) |  |  |  |  |
  CYCLE 4 DAY 1 0 h: number analyzed (Participants) | 1 | 2 | 3 | 3 | 2 | 3 | 5 | 5 | 6 | 5 | 1 | 3 | 1 | 2 | 2 | 15 | 2 | 0 | 3 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0
  CYCLE 4 DAY 1 0 h | 3420 (NA) — No measure of variation/dispersion for a single data value | 4593 (24.0) | 7169 (37.3) | 20703 (32.1) | 26090 (13.0) | 358 (95.8) | 2095 (96.5) | 5108 (71.4) | 20800 (43.7) | 47108 (45.2) | 1080 (NA) — No measure of variation/dispersion for a single data value | 1971 (51.3) | 5140 (NA) — No measure of variation/dispersion for a single data value | 12649 (78.3) | 32150 (0.660) | 7252 (43.4) | 1466 (72.4) |  | 754 (48.1) |  |  | 5461 (26.4) |  |  |  |  |
  CYCLE 4 DAY 29 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
  CYCLE 4 DAY 29 0 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1856 (75.1) |  |  |  |  |
  CYCLE 4 DAY 15 336 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
  CYCLE 4 DAY 15 336 h |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 2130 (69.4) |  |  |  |  |
  CYCLE 5 DAY 1 0 h: number analyzed (Participants) | 0 | 1 | 2 | 1 | 1 | 3 | 3 | 7 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 11 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 5 DAY 1 0 h |  | 6600 (NA) — No measure of variation/dispersion for a single data value | 13491 (36.0) | 13300 (NA) — No measure of variation/dispersion for a single data value | 35200 (NA) — No measure of variation/dispersion for a single data value | 386 (84.8) | 1301 (100) | 7468 (55.1) | 26813 (52.7) | 90700 (NA) — No measure of variation/dispersion for a single data value |  |  |  |  |  | 9811 (37.3) | 1671 (63.5) |  |  |  |  |  |  |  |  |  |
  CYCLE 5 DAY 1 504 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 5 DAY 1 504 h |  |  |  |  |  |  |  |  |  |  |  | 2527 (67.6) |  |  | 18771 (45.0) |  |  |  | 1262 (10.2) |  |  |  |  |  |  |  |
  CYCLE 6 DAY 1 0 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  CYCLE 6 DAY 1 0 h |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 604 (138) |  |  |  |  |
  CYCLE 6 DAY 1 672 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 6 DAY 1 672 h |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 62.5 (NA) — No measure of variation/dispersion for a single data value |  |  |  |  |  |  |  |  |  |
  CYCLE 7 DAY 1 0 h: number analyzed (Participants) | 0 | 1 | 2 | 2 | 0 | 1 | 3 | 4 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 7 DAY 1 0 h |  | 5390 (NA) — No measure of variation/dispersion for a single data value | 10217 (45.8) | 22073 (60.3) |  | 946 (NA) — No measure of variation/dispersion for a single data value | 4777 (75.6) | 12527 (58.8) | 32753 (53.9) | 76970 (33.0) |  |  |  |  |  | 11471 (38.5) |  |  |  |  |  |  |  |  |  |  |
  CYCLE 9 DAY 1 0 h: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 9 DAY 1 0 h |  |  | 6300 (NA) — No measure of variation/dispersion for a single data value | 31300 (NA) — No measure of variation/dispersion for a single data value |  |  | 6397 (50.5) | 13536 (105) | 29902 (30.0) | 106710 (40.9) |  |  |  |  |  | 12905 (42.4) |  |  | 579 (NA) — No measure of variation/dispersion for a single data value |  |  |  |  |  |  |  |
  CYCLE 10 DAY 1 0 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 10 DAY 1 0 h |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 29100 (NA) — No measure of variation/dispersion for a single data value |  |  |  |  |  |  |  |  |  |  |  |
  CYCLE 10 DAY 1 336 h: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 10 DAY 1 336 h |  |  | 6470 (NA) — No measure of variation/dispersion for a single data value | 33600 (NA) — No measure of variation/dispersion for a single data value |  | 1190 (NA) — No measure of variation/dispersion for a single data value | 8264 (44.0) | 5686 (78.2) | 28988 (33.9) | 131520 (70.3) |  |  |  |  |  | 13400 (26.3) |  |  |  |  |  |  |  |  |  |  |
  CYCLE 17 DAY 1 0 h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CYCLE 17 DAY 1 0 h |  |  |  |  |  |  |  |  | 48500 (NA) — No measure of variation/dispersion for a single data value |  |  |  |  |  |  | 16600 (NA) — No measure of variation/dispersion for a single data value |  |  |  |  |  |  |  |  |  |  |

24. Secondary Outcome: Frequency of Positive Anti-Drug Antibodies (ADA) to BMS-986178
Description: The number of participants with positive anti-drug antibodies (ADA) is assessed to characterize the immunogenicity of BMS-986178 administered alone or in combination with nivolumab and/or ipilimumab. ADA Positive: A participant with at least one ADA-positive sample relative to baseline (ADA negative at baseline or ADA titer to be at least 4-fold or greater (>=) than baseline positive titer) at any time after initiation of treatment.
Time Frame: Cycle 1-6 timepoints can include (Pre-dose, 696 hours post dose)
Population: All BMS 986178 Treated Participants with Baseline and at Least One Post-baseline ADA Assessment (Parts 1-9)
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 1 | 2 | 3 | 3 | 3 | 6 | 6 | 6 | 7 | 5 | 2 | 5 | 6 | 7 | 6 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0
Participants | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 3 | 1 | 0 | 1 | 3 | 1 | 4 | 2 |  | 1 |  |  |  |  | 0 | 0 | 0 |  |

25. Secondary Outcome: Frequency of Positive Anti-Drug Antibodies (ADA) to Nivolumab
Description: The number of participants with positive anti-drug antibodies (ADA) is assessed to characterize the immunogenicity of Nivolumab administered with BMS-986178 ADA Positive: A participant with at least one ADA-positive sample relative to baseline (ADA negative at baseline or ADA titer to be at least 4-fold or greater (>=) than baseline positive titer) at any time after initiation of treatment.
Time Frame: Cycle 1-6 timepoints can include (Pre-dose, 336, 696 hours post dose)
Population: All BMS 986178 Treated Participants with Baseline and at Least One Post-baseline ADA Assessment (Parts 1-9)
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 5 | 7 | 8 | 8 | 6 | 17 | 9 | 5 | 1 | 5 | 9 | 0 | 1 | 0 | 1 | 0
Participants | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 1 |  | 1 |  | 0 |

26. Secondary Outcome: Frequency of Positive Anti-Drug Antibodies (ADA) to Ipilimumab.
Description: The number of participants with positive anti-drug antibodies (ADA) is assessed to characterize the immunogenicity of Ipilimumab administered with BMS-986178 ADA Positive: A participant with at least one ADA-positive sample relative to baseline (ADA negative at baseline or ADA titer to be at least 4-fold or greater (>=) than baseline positive titer) at any time after initiation of treatment.
Time Frame: Cycle 1-6 timepoints can include (Pre-dose, 696 hours post dose)
Population: All BMS 986178 Treated Participants with Baseline and at Least One Post-baseline ADA Assessment (Parts 1-9)
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC)
Number analyzed (Participants) | 4 | 5 | 7 | 7 | 6 | 6 | 6 | 1 | 5 | 9
Participants | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: The Number of Participants Showing a Change in Soluble OX40 and Peripheral OX40 Receptor Occupancy Pharmacodynamic Biomarkers in Part 8
Description: The Number of Participants Showing a Change in Soluble OX40 and Peripheral OX40 Receptor Occupancy Pharmacodynamic Biomarkers in Part 8. A threshold of 80% receptor occupancy following treatment was applied.
Time Frame: Cycle 1-6 timepoints can include (Pre-dose, 24, 168, 336, 672, 1848 hours post dose)
Population: All treated participants with Pharmacodynamic biomarker assessments (Part 8)
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W
Number analyzed (Participants) | 2 | 2 | 2 | 2
Participants
  Soluble OX40: number analyzed (Participants) | 0 | 0 | 0 | 0
  Peripheral OX40 receptor occupancy (CD4+ T cells): number analyzed (Participants) | 1 | 2 | 1 | 1
  Peripheral OX40 receptor occupancy (CD4+ T cells) | 1 | 2 | 1 | 0
  Peripheral OX40 receptor occupancy (Tregs): number analyzed (Participants) | 1 | 2 | 1 | 1
  Peripheral OX40 receptor occupancy (Tregs) | 1 | 1 | 1 | 0

28. Secondary Outcome: Tumor Pharmacodynamics of BMS-986178 in Combination With Nivolumab or Nivolumab Monotherapy in Part 8
Description: Tumor pharmacodynamics of BMS-986178 in combination with nivolumab or nivolumab monotherapy
Time Frame: Screening, cycle 1-2 timepoints can include (Pre-dose, 336, 1848 hours post dose)
Population: Tumor pharmacodynamic readouts not possible due to only 1 matched pair
Arm/Group | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W
Number analyzed (Participants) | 0 | 0 | 0 | 0

29. Secondary Outcome: The Number of Participants With Sustained T Cell Expansion With DPV-001 in Combination With Nivolumab or Nivolumab Monotherapy in Part 9
Description: The number of participants with Sustained T Cell Expansion with DPV-001 in Combination with Nivolumab or Nivolumab Monotherapy was assessed to show a change in pharmacodynamics biomarkers
Time Frame: Cycle 1-6 timepoints can include (Pre-dose, 24, 168, 336, 672, 1848 hours post dose)
Population: All treated participants with available biomarker data (Part 9)
Arm/Group | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first dose to 100 days post last dose (up to 2.5 years) All Cause Mortality from first dose to study completion (up to approximately 4 years 5 months)
Arm/Group | Escalation Part 1: BMS 20 mg Q2W | Escalation Part 1: BMS 40 mg Q2W | Escalation Part 1: BMS 80 mg Q2W | Escalation Part 1: BMS 160 mg Q2W | Escalation Part 1: BMS 320 mg Q2W | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine
All-Cause Mortality (participants affected / at risk) | 4/4 | 4/4 | 3/4 | 4/4 | 4/4 | 3/7 | 7/8 | 11/12 | 6/8 | 6/8 | 4/4 | 9/10 | 7/7 | 8/8 | 2/6 | 16/18 | 11/12 | 3/6 | 3/7 | 0/1 | 5/6 | 4/9 | 2/2 | 2/2 | 1/2 | 1/2 | 1/1
Serious Adverse Events (participants affected / at risk) | 3/4 | 4/4 | 2/4 | 3/4 | 3/4 | 3/7 | 6/8 | 7/12 | 4/8 | 5/8 | 2/4 | 6/10 | 6/7 | 5/8 | 2/6 | 11/18 | 7/12 | 4/6 | 4/7 | 1/1 | 6/6 | 5/9 | 0/2 | 1/2 | 1/2 | 1/2 | 1/1
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4 | 3/4 | 4/4 | 7/7 | 8/8 | 12/12 | 6/8 | 8/8 | 4/4 | 10/10 | 7/7 | 8/8 | 6/6 | 18/18 | 11/12 | 6/6 | 5/7 | 1/1 | 6/6 | 9/9 | 2/2 | 2/2 | 2/2 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escalation Part 1: BMS 20 mg Q2W (N=4) | Escalation Part 1: BMS 40 mg Q2W (N=4) | Escalation Part 1: BMS 80 mg Q2W (N=4) | Escalation Part 1: BMS 160 mg Q2W (N=4) | Escalation Part 1: BMS 320 mg Q2W (N=4) | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W (N=7) | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W (N=8) | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W (N=12) | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W (N=8) | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W (N=8) | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W (N=4) | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W (N=10) | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W (N=7) | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W (N=8) | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W (N=6) | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) (N=18) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W (N=12) | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W (N=6) | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) (N=7) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) (N=1) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) (N=6) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) (N=9) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W (N=2) | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W (N=2) | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W (N=2) | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W (N=2) | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected fistula (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 2 | 2 | 1 | 1 | 3 | 5 | 1 | 4 | 2 | 5 | 5 | 4 | 1 | 6 | 1 | 1 | 2 | 0 | 4 | 1 | 0 | 0 | 0 | 1 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bell's palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Secondary cerebellar degeneration (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Escalation Part 1: BMS 20 mg Q2W (N=4) | Escalation Part 1: BMS 40 mg Q2W (N=4) | Escalation Part 1: BMS 80 mg Q2W (N=4) | Escalation Part 1: BMS 160 mg Q2W (N=4) | Escalation Part 1: BMS 320 mg Q2W (N=4) | Escalation Part 2 BMS 20 mg + Nivo 240 mg Q2W (N=7) | Escalation Part 2: BMS 40 mg + Nivo 240 mg Q2W (N=8) | Escalation Part 2: BMS 80 mg + Nivo 240 mg Q2W (N=12) | Escalation Part 2: BMS 160 mg + Nivo 240 mg Q2W (N=8) | Escalation Part 2: BMS 320 mg + Nivo 240 mg Q2W (N=8) | Escalation Part 3: BMS 20 mg + Ipi 1 mg/kg Q3W (N=4) | Escalation Part 3: BMS 40 mg + Ipi 1 mg/kg Q3W (N=10) | Escalation Part 3: BMS 80 mg + Ipi 1 mg/kg Q3W (N=7) | Escalation Part 3: BMS 160 mg + Ipi 1 mg/kg Q3W (N=8) | Escalation Part 3: BMS 320 mg + Ipi 1 mg/kg Q3W (N=6) | Expansion Part 2C: BMS 80 mg + Nivo 240 mg Q2W (BDC) (N=18) | Schedule and Dose Exploration Part 4: BMS 80 mg + Nivo 480 mg Q4W (N=12) | Schedule and Dose Exploration Part 5: BMS 80 mg + Ipi 3 mg/kg Q3W (N=6) | Safety Part 6A: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) (N=7) | Expansion Part 6B: BMS 40 mg + Nivo 240 mg + Ipi 1 mg/kg Q3W / BMS 40 mg + Nivo 480 mg Q4W (RCC) (N=1) | Safety Cohort Part 7A: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) (N=6) | Expansion Part 7B: BMS 40mg Q2W + Nivo 240 mg Q2W + Ipi 1 mg/kg Q6W (NSCLC) (N=9) | Schedule and Dose Exploration Part 8: Cohort 1- BMS 20 mg Q12W + Nivo 480 mg Q4W (N=2) | Schedule and Dose Exploration Part 8: Cohort 2- BMS 40 mg Q12W + Nivo 480 mg Q4W (N=2) | Schedule and Dose Exploration Part 8: Cohort 3- BMS 80 mg Q12W + Nivo 480 mg Q4W (N=2) | Schedule and Dose Exploration Part 8: Cohort 4- Nivo 480 mg Q4W (N=2) | Exploration Part 9 Cohort 1: BMS 40 mg Q4W + Nivo 480 mg Q4W + DRibble Vaccine (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 0 | 3 | 4 | 2 | 1 | 1 | 0 | 3 | 2 | 3 | 2 | 8 | 5 | 2 | 2 | 0 | 1 | 3 | 0 | 1 | 0 | 2 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid rash (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 2 | 2 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 0 | 1 | 2 | 4 | 3 | 1 | 1 | 5 | 0 | 0 | 3 | 3 | 2 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 2 | 2 | 4 | 2 | 1 | 3 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 1 | 2 | 1 | 3 | 2 | 2 | 1 | 2 | 2 | 2 | 0 | 0 | 3 | 4 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 1 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Early satiety (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 5 | 4 | 0 | 2 | 1 | 2 | 2 | 7 | 3 | 4 | 3 | 1 | 1 | 4 | 0 | 1 | 1 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injury associated with device (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 5 | 0 | 2 | 1 | 4 | 0 | 1 | 0 | 4 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temperature regulation disorder (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cryptosporidiosis infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sputum purulent (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular access site occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ammonia increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood chloride increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactic acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carbon dioxide decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lymph node palpable (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Serum ferritin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine protein/creatinine ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 0 | 2 | 2 | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 7 | 1 | 2 | 0 | 3 | 2 | 3 | 1 | 3 | 0 | 1 | 3 | 2 | 1 | 1 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 2 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight bearing difficulty (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bell's palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Secondary cerebellar degeneration (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 1 | 4 | 1 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 4 | 2 | 2 | 1 | 1 | 5 | 0 | 0 | 1 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Autoimmune dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 2 | 2 | 3 | 3 | 1 | 0 | 1 | 5 | 0 | 0 | 2 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism venous (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT02737475/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT02737475/SAP_001.pdf